CLINICAL TRIAL: NCT00350909
Title: Brief Intervention for Drug Abusing Students
Brief Title: Brief Intervention for Drug Abusing Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Ken Winters, ph.D., Dept. of Psychiatry, University of Minnesota
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0308S51681
Record Dates: First submitted 2006-07-07; First posted 2006-07-11 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Drug Abuse
Keywords: drug abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Crisis Intervention; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): One arm was a 2-session brief intervention with both sessions involving only the adolescent. Each session was a 60 minute individual session with the counselor.
  Interventions: Behavioral: brief intervention (cognitive-behavioral therapy)
- 2 (Active Comparator): The other arm was a 3-session brief intervention, with 2 sessions involving the adolescent and one session with the parent. Each of these individual sessions were 60 minutes.
  Interventions: Behavioral: brief intervention (cognitive-behavioral therapy)

INTERVENTIONS:
Behavioral: brief intervention (cognitive-behavioral therapy) — Consists of 60 minute individual sessions delivered with a therapist using a motivational interviewing (MI) style. Session 1 focuses on eliciting information about the students' substance use and related consequences based on the assessment, their perception of level of willingness to change, examining the cause and benefits of change using the decisional balance exercise, and discussing what goals for change the student would like to select and pursue. Session 2 reviewed the students' progress with the agreed upon goals, identifying high risk situations associated with clients difficulty in achieving the goals, discussing strategies to address barriers toward goal attainment, reviewing where the client is in the stage of change process, and negotiating either the continuation of goals or advancing to more ambitious goals of substance use reduction. Session 3 involved delivering the same MI interviewing style to the primary parent or guardian (student is not present).
  Other Names: cognitive-behavioral therapy- motivational interviewing

SUMMARY:
The purpose of this clinical trail is to evaluate the efficacy of a brief, cognitive-behavioral therapeutic intervention for adolescents reporting mild or moderate drug abuse (MMDA). This school-based initiative employs a collaborative effort between the University of Minnesota researchers and the St. Paul Public Schools. This intervention aims to reduce post-treatment drug use behaviors and enhance drug-use resistant cognitions and problem-solving skills.

DETAILED DESCRIPTION:
The purpose of this clinical trail is to evaluate the efficacy of a brief, cognitive-behavioral therapeutic intervention for adolescents reporting mild or moderate drug abuse (MMDA). This school-based initiative employs a collaborative effort between the University of Minnesota researchers and the St. Paul Public Schools. This intervention aims to reduce post-treatment drug use behaviors and enhance drug-use resistant cognitions and problem-solving skills.

Specifically, we propose a randomized clinical trial to evaluate the efficacy of a cognitive-behavioral therapy on key process and outcome dimensions among school-based youth with mild-to-moderate drug abuse (MMDA). The experimental treatment is designated Brief Cognitive Behavioral Intervention (BCBI) given its theoretical foundation in stage of change theory used to coordinate modules on Rational-Emotive Therapy and Problem Solving Therapy. BCBI will be compared against a second experimental treatment that consists of BCBI and a single parent session (BCBI+P) and an assessment only condition (control). The importance of clarifying mechanisms in drug treatment research will be explored with respect to a limited number of treatment and individual factors that have emerged as promising mediating and moderating factors, such as cognitive and problem solving factors, parenting practices, and peer group influences.

ELIGIBILITY:
Inclusion Criteria:

1. student at a local school
2. meets DSM-IV criteria for a substance abuse disorder for at least one drug
3. student and parent both agree to participate in the intervention study

Exclusion Criteria:

1. meets criteria for at least one DSM-IV substance dependence disorder
2. meets criteria for a psychotic disorder or a learning disability

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2005-09; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Drug use frequency and quantity at 1-, 3- and 12-months post-intervention. | 1 year post treatment

SECONDARY OUTCOMES:
HIV and sexual risk behaviors at the same time period. | 1 year post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ken C Winters, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Piehler TF, Winters KC. Decision-making style and response to parental involvement in brief interventions for adolescent substance use. J Fam Psychol. 2017 Apr;31(3):336-346. doi: 10.1037/fam0000266. Epub 2016 Dec 8. PMID 27929312